CLINICAL TRIAL: NCT07174063
Title: An Open-label, Single-arm Study to Evaluate the Safety, Tolerability and Pharmacokinetics of JSB462 (Luxdegalutamide) in Japanese Patients With Metastatic Prostate Cancer
Brief Title: A Phase I Study of JSB462 (Luxdegalutamide) in Japanese Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJSB462A11101
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Cancer (mCRPC)
Keywords: metastatic prostate cancer (mCRPC); JSB462; luxdegalutamide; open-label
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive JSB462 orally, daily and continuously (100 mg or 300 mg QD).
  Interventions: Drug: JSB462

INTERVENTIONS:
Drug: JSB462 — 300 mg or 100 mg once a day (QD) with food

SUMMARY:
This Phase I study aims to evaluate the safety, tolerability and PK of JSB462 in Japanese patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
Participants will receive JSB462 at the starting dose of 300 mg QD to evaluate its safety, tolerability and PK. Any Adverse Events (AEs) and Dose Limiting Toxicities (DLTs) will be assessed. DLTs will be evaluated in the first (28-day) cycle. If 300 mg once a day (QD) is considered intolerable by investigators and Novartis study personnel during dose evaluation meeting, the tolerability of 100 mg QD dose level cohort may be assessed.

Study treatment will be administered until disease progression (per PCWG3-modified RECIST v1.1 assessed by the investigator), unacceptable toxicity, death, withdrawal of consent, lost to follow-up or investigator's decision.

The End of Treatment Visit and the Safety Follow-up Visit will be performed within 7 days and 30 days from the last dose of JSB462, respectively. If participants discontinue study treatment for reasons other than disease progression (per PCWG3-modified RECIST v1.1 assessed by the investigator), death, lost to follow-up, or withdrawal of consent, then tumor assessments should continue to be performed in the Efficacy Follow-up Visit according to the planned schedule until disease progression (per PCWG3-modified RECIST v1.1 assessed by the investigator), death, withdrawal of consent or lost to follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult male patients with histologically or cytologically confirmed and documented adenocarcinoma of the prostate.
* At least 1 bone or visceral metastatic lesion (according to local radiology assessment by the investigator) present on baseline CT, MRI, or bone scan imaging obtained ≤28 days prior to enrollment. Lymph nodes as only site of metastases are not allowed.
* Patients with prostate cancer must have failed or refused available standard therapies, be intolerant or ineligible to receive such therapy, or for whom no standard therapy exists.
* Patients must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L). Ongoing ADT (as defined by prior orchiectomy and/or ongoing GnRH analog/antagonist) is allowed prior to enrollment.
* Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1.

Key Exclusion Criteria:

* Patients with CNS metastases.
* Patients with any other active malignancy other than prostate cancer. Exceptions to this criterion include the following: malignancies that were treated curatively at least 3 years before starting study treatment which have not recurred; basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative local therapy or other tumors that will not affect life expectancy.

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-06-18 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) during the first cycle of treatment | Up to 28 days
  A dose-limiting toxicity (DLT) is defined as a treatment-related adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness/injury, or concomitant medications that occurs within the first 28 days of treatment with JSB462 and meets any of the criteria specified in the protocol. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for all grading. For the purpose of dose regimen decisions, DLTs will be considered.
Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, an average of approximately 18 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Number of Participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 18 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by means of descriptive statistics.
Dose Intensity | From date of randomization till 30 days safety fup, assessed up to approximately 18 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized by means of descriptive statistics.
Plasma concentrations of JSB462 and its metabolite ARV-767 | Cycle 1: Days 1 & 21 (0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Days 2 & 22 (0 hour). Cycles 2-6: Day 1 (0 hour). End of Treatment Visit (EOT): within 7 days from the last dose of JSB462. 1 cycle = 28 days.
  JSB462 pharmacokinetic (PK) samples will be obtained and evaluated to assess single dose and steady-state plasma Pharmacokinetic (PK) of JSB462 and its metabolite ARV-767 and summarized using descriptive statistics.
AUC of JSB462 | Cycle 1: Days 1 & 21 (0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Days 2 & 22 (0 hour). Cycles 2-6: Day 1 (0 hour). End of Treatment Visit (EOT): within 7 days from the last dose of JSB462. 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) and Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) will be listed and summarized using descriptive statistics.
Cmax of JSB462 | Cycle 1: Days 1 & 21 (0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Days 2 & 22 (0 hour). Cycles 2-6: Day 1 (0 hour). End of Treatment Visit (EOT): within 7 days from the last dose of JSB462. 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Tmax of JSB462 | Cycle 1: Days 1 & 21 (0 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Days 2 & 22 (0 hour). Cycles 2-6: Day 1 (0 hour). End of Treatment Visit (EOT): within 7 days from the last dose of JSB462. 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Kobe

IPD SHARING:
Plan to Share IPD: No